CLINICAL TRIAL: NCT05257200
Title: Intestinal Permeability in Patients With Liver Fibrosis and NASH Progression Undergoing Bariatric-metabolic Surgery
Brief Title: Gut Permeability and Bariatric-metabolic Surgery
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Prager, Professor of Bariatric Surgery, Medical University of Vienna
Other Study IDs: 2180/2020
Record Dates: First submitted 2022-01-10; First posted 2022-02-25 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Bariatric Surgery Candidate; Intestinal Permeability
Keywords: liver fibrosis; NAFLD; One Anastomosis Gastric Bypass; Roux-en-Y Gastric Bypass; Gut-liver axis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Increased intestinal permeability and dysbiosis have been causally associated with NAFLD and NASH progression. However, to date, there are no systematic studies, on the effect of bariatric-metabolic surgery on intestinal permeability and dysbiosis in the context of NAFLD development.

DETAILED DESCRIPTION:
Morbid obesity is associated with non-alcoholic fatty liver disease (NAFLD) in 80-90% of patients, and non-alcoholic steatohepatitis (NASH) occurs in up to 60% of patients. If left untreated, the disease can progress to liver fibrosis, cirrhosis, or hepatocellular carcinoma. Weight loss of >10% of body weight is the most effective treatment for NAFLD, and bariatric metabolic surgery plays an effective role in achieving long-term weight loss. About 80% of patients achieve improvement or reversal of NAFLD after bariatric-metabolic surgery. However, clinical and histological progression of liver disease may occur in about 20% of patients, despite weight the loss. Increased intestinal permeability and dysbiosis have been causally associated with NAFLD and NASH progression. However, to date, there are no systematic studies, on intestinal permeability and dysbiosis after bariatric-metabolic surgery.

Research questions

* To investigate the changes in intestinal permeability after bariatric-metabolic surgery.
* To investigate the differences in intestinal permeability at the time of surgery and 1 year after surgery between patients with liver fibrosis grades F≤1 and F≥2 (low-grade fibrosis vs advanced fibrosis).
* To investigate differences between patients with and without liver fibrosis progression using parameters for metabolic endotoxemia, intestinal permeability, and dysbiosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with morbid obesity undergoing bariatric metabolic surgery according to the IFSO criteria,
* Willingness to attend all follow-up visits
* Written consent

Exclusion Criteria:

* other liver disease than NAFLD
* presence of IBD, acute pancreatitis, amyotrophic lateral sclerosis, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our patients about 80% have NAFLD, about 50-60% are diagnosed with NASH. Furthermore, we know from our obese patient cohort, that 26% are diagnosed with fibrosis grade 2 or higher. Only patients that are scheduled for weight loss surgery will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Intestinal Permeability improves with significant weight loss after bariatric metabolic surgery | 12 months observation period
  At the time of surgery and 12 months after surgery a multisugar (lactulose-mannitol) test will be performed, stool and blood samples will be taken. During surgery small bowel biopsies and liver biopsies will be taken. For the 12 months visit noninvasive fibrosis markers will be calculated, transient elastography will be performed and compared to the results from the intestinal permeability assays.
  Analysis will be performed on anonymized data only. A list cross-linking the patient number to the name will be kept secure and is only available to the principal researcher. Written informed consent will be kept for 15 years. Missing data will not be imputed but reported upon in the results.
Refractory fibrosis or fibrosis progression after bariatric surgery is associated with persistent intestinal permeability | 12 months observation period
  At the time of surgery and 12 months after surgery a multisugar (lactulose-mannitol) test will be performed, stool and blood samples will be taken. During surgery small bowel biopsies and liver biopsies will be taken. For the 12 months visit noninvasive fibrosis markers will be calculated, transient elastography will be performed and compared to the results from the intestinal permeability assays.
  Analysis will be performed on anonymized data only. A list cross-linking the patient number to the name will be kept secure and is only available to the principal researcher. Written informed consent will be kept for 15 years. Missing data will not be imputed but reported upon in the results.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria